CLINICAL TRIAL: NCT03077607
Title: A PHASE 1 OPEN-LABEL, TWO-ARM,DRUG-DRUG INTERACTION STUDY TO EVALUATE THE EFFECT OF ITRACONAZOLE AND RIFAMPIN ON THE PHARMACOKINETICS OF TALAZOPARIB IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Evaluate the Effect of Itraconazole and Rifampin on the Pharmacokinetics of Talazoparib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-04; C3441004 (Other: Alias Study Number); 2016-001813-26 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-03-13 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — talazoparib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Subjects will receive a 0.5 mg talazoparib and 100 mg itraconazole.
  Interventions: Drug: Talazoparib; Drug: Itraconazole
- Arm B (Experimental): Subjects will receive 1 mg talazoparib and 600 mg rifampin.
  Interventions: Drug: Talazoparib; Drug: Rifampin

INTERVENTIONS:
Drug: Talazoparib — Arm A: 0.5 mg oral dose Arm B: 1 mg oral dose
Drug: Itraconazole — 100 mg oral dose
  Arms: Arm A
Drug: Rifampin — 600 mg oral dose
  Arms: Arm B

SUMMARY:
This is a study in patients with advanced solid tumors for the investigation of P-gp inhibition and induction on the PK of talazoparib.

DETAILED DESCRIPTION:
Subjects participating in this study with no clinically significant toxicities and no disease progression may be eligible to continue treatment on a separate extension protocol (MDV3800-13).

ELIGIBILITY:
Inclusion Criteria:

1. Arm A: At least 18 years of age and <65 years of age (at the time point of consent) and willing and able to provide informed consent. Arm B: At least 18 years of age (at the time point of consent) and willing and able to provide informed consent.
2. Histologically confirmed advanced solid tumor (limited to platinum-resistant ovarian carcinoma, cervical adenocarcinoma, small cell lung carcinoma or triple-negative breast cancer) judged by the Investigator to not be appropriate for standard therapy.
3. ECOG performance status ≤ 2 at screening and at time of enrollment.
4. Expected life expectancy of ≥ 3 months.
5. Able to swallow the study drug and comply with study requirements.
6. Female subjects may be enrolled if they are considered not of childbearing potential, or who are post-menopausal, or are of childbearing potential using a highly effective form of contraceptive, and female subjects should not donate eggs from the time point of investigational medicinal product (IMP) administration until at least 45 days thereafter.
7. Males with partners of childbearing potential may be enrolled if they use a condom when having sex with a pregnant woman or with a woman of childbearing potential, and do not donate sperm from the time point of study drug administration until at least 105 days thereafter, and males should not donate sperm from the time point of study drug administration until at least 105 days thereafter.
8. Female subjects must not be breastfeeding at screening and during the study participation until 45 days after the last dose of the study drug.
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Treatment within 14 days or 5 half lives prior to dosing with any type of systemic anticancer therapy or any investigational agent, whichever is longer
2. Major surgery within 8 weeks before screening.
3. Serious accompanying disorder or impaired organ function.
4. Symptomatic or impending spinal cord compression or cauda equina syndrome.
5. Non-healing wound, ulcer, or bone fracture, not including a pathological bone fracture caused by a pre-existent pathological bone lesion.
6. Known myelodysplastic syndrome.
7. Subjects with the following serologies should be excluded: HBsAg+ or anti-HBc+;HCV+; HIV+.
8. Serious or unstable medical condition that interferes with ability to tolerate treatment or assessments associated with the protocol.
9. Gastrointestinal disorder affecting absorption.
10. Known hypersensitivity to any of the talazoparib capsule components.
11. Any condition or reason that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator or Sponsor (e.g. non-compliance, excessive alcohol consumption, intake of drugs of abuse unless these drugs are medically indicated [e.g. opiates for pain relief].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- PRA Magyarorszag Kft, Fazis I-es Klinikai Farmakologiai Vizsgalohely, Budapest, Hungary
- ARENSIA Exploratory Medicine Phase I Unit, PMSI Institute of Oncology, Chisinau, Moldova
- Szpital LUX MED, Warsaw, Poland
- Russia (3):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - "BioEq" LLC, Saint Petersburg
  - State budget healthcare institution of Yaroslavl region "Regional clinical oncology hospital", Yaroslavl

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Elmeliegy M, Lang I, Smolyarchuk EA, Chung CH, Plotka A, Shi H, Wang D. Evaluation of the effect of P-glycoprotein inhibition and induction on talazoparib disposition in patients with advanced solid tumours. Br J Clin Pharmacol. 2020 Apr;86(4):771-778. doi: 10.1111/bcp.14178. Epub 2020 Jan 7. PMID 31770456
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-04

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted in 4 countries from 07-Nov-2016 to 18 Dec 2017.
Groups:
- A: Talazoparib 0.5 mg + Itraconazole 100 mg BID: Participants received a single oral dose of talazoparib 0.5 milligram (mg) on Day 1, which was followed by a wash out of 14 days in Period 1. Then in Period 2 participants received oral dose of itraconazole 200 mg (100 mg twice daily [BID]) from Day 16 to Day 36 and a single oral dose of talazoparib 0.5 mg on Day 23. Participants were followed up to 23 days after last dose of study drug.
- B: Talazoparib 1 mg + Rifampin 600 mg QD: Participants received a single oral dose of talazoparib 1.0 mg on Day 1, which was followed by a wash out of 14 days in Period 1. Then in Period 2 participants received oral dose of rifampin 600 mg once daily (QD) from Day 16 to Day 38 and a single oral dose of talazoparib 1.0 mg on Day 25. Participants were followed up to 23 days after last dose of study drug.
Period: Period 1 (15 Days)
Arm/Group | A: Talazoparib 0.5 mg + Itraconazole 100 mg BID | B: Talazoparib 1 mg + Rifampin 600 mg QD
Started | 19 | 17
Treated (With Any Study Drug) | 19 | 17
Received Talazoparib | 19 | 17
Completed | 17 | 17
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Period: Period 2 (Arm A:21 Days; Arm B:23 Days)
Arm/Group | A: Talazoparib 0.5 mg + Itraconazole 100 mg BID | B: Talazoparib 1 mg + Rifampin 600 mg QD
Started | 17 | 17
Treated (With Any Study Drug) | 17 | 17
Received Talazoparib | 15 | 15
Completed | 14 | 15
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of talazoparib.
Groups:
- A: Talazoparib 0.5 mg + Itraconazole 100 mg BID: Participants received a single oral dose of talazoparib 0.5 mg on Day 1, which was followed by a wash out of 14 days in Period 1. Then in Period 2 participants received oral dose of itraconazole 200 mg (100 mg BID) from Day 16 to Day 36 and a single oral dose of talazoparib 0.5 mg on Day 23. Participants were followed up to 23 days after last dose of study drug.
- B: Talazoparib 1 mg + Rifampin 600 mg QD: Participants received a single oral dose of talazoparib 1.0 mg on Day 1, which was followed by a wash out of 14 days in Period 1. Then in Period 2 participants received oral dose of rifampin 600 mg QD from Day 16 to Day 38 and a single oral dose of talazoparib 1.0 mg on Day 25. Participants were followed up to 23 days after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | A: Talazoparib 0.5 mg + Itraconazole 100 mg BID | B: Talazoparib 1 mg + Rifampin 600 mg QD | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 4 | 23
  >=65 years | 0 | 13 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib: Alone and in Combination With Itraconazole
Description: T1= Time frame for "Talazoparib 0.5 mg Alone" and T2= time frame for "Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID".
Time Frame: T1=Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 and 336 hours post Talazoparib dose on Day 1; T2=Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 and 336 hours post Talazoparib dose on Day 23
Population: Pharmacokinetic (PK) analysis population included all participants who enrolled, treated and had at least 1 of the talazoparib PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Groups:
- Talazoparib 0.5 mg Alone: Participant received a single oral dose of talazoparib 0.5 mg on Day 1 followed by washout of 14 days in Period 1.
- Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID: Participants received a single oral dose of talazoparib 0.5 mg on Day 23 and oral dose of itraconazole 200 mg (100 mg BID) from Day 23 onwards to Day 36 in Period 2.
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 19 | 15
Picogram per milliliter (pg/mL) | 2092.00 (50) | 2936.82 (56)
Statistical Analysis 1: Comparison: Talazoparib 0.5 mg Alone vs Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID; Confidence interval (CI): 90 percent (%) CI on geometric least squares (LS) mean ratio (Test/Reference), test is talazoparib in combination with itraconazole and reference is talazoparib alone. Statistical data was calculated by using analysis of variance (ANOVA); Test type: Equivalence — Sample size of 15 participants was selected based on the estimated within participant % coefficient of variation (CV) of 42% and precision/half width of 90% CI for Test Reference comparison on log scale of 0.259; Geometric LS Mean Ratio = 139.92, 90% CI 2-sided [113.26 to 172.87]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of Talazoparib: Alone and in Combination With Itraconazole
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK analysis population included all participants who enrolled, treated and had at least 1 of the talazoparib PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter (hr*pg/mL)
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 19 | 15
Hour*picogram per milliliter (hr*pg/mL) | 98532.30 (38) | 145944.59 (38)
Statistical Analysis 1: Comparison: Talazoparib 0.5 mg Alone vs Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID; CI: 90% CI on geometric LS mean ratio (Test/Reference), test is talazoparib in combination with itraconazole and reference is talazoparib alone. Statistical data was calculated by using ANOVA; Test type: Equivalence — Sample size of 15 participants was selected based on the estimated within participant %CV of 42% and precision/half width of 90% CI for Test Reference comparison on log scale of 0.259; Geometric LS Mean Ratio = 150.71, 90% CI 2-sided [136.47 to 166.43]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinity (AUC0-inf) of Talazoparib: Alone and in Combination With Itraconazole
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK analysis population included all participants who enrolled, treated and had at least 1 of the talazoparib PK parameters. Here, "Overall number of participants analyzed" (N) signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 18 | 12
hr*pg/mL | 109762.10 (42) | 151919.63 (36)
Statistical Analysis 1: Comparison: Talazoparib 0.5 mg Alone vs Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 156.24, 90% CI 2-sided [137.58 to 177.42]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib: Alone and in Combination With Rifampin
Description: T3= Time frame for "Talazoparib 1.0 mg Alone" and T4= time frame for "Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD".
Time Frame: T3=Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 and 336 hours post Talazoparib dose on Day 1; T4=Predose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264 and 336 hours post Talazoparib dose on Day 25
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Talazoparib 1.0 mg Alone: Participant received a single oral dose of talazoparib 1.0 mg on Day 1 followed by washout of 14 days in Period 1.
- Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD: Participants received a single oral dose of talazoparib 1.0 mg on Day 25 and oral dose of rifampin 600 mg QD from Day 25 onwards to Day 38 in Period 2.
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 15
pg/mL | 6007.01 (53) | 8336.83 (71)
Statistical Analysis 1: Comparison: Talazoparib 1.0 mg Alone vs Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD; CI: 90% CI on geometric LS mean ratio (Test/Reference), test is talazoparib in combination with rifampin and reference is talazoparib alone. Statistical data was calculated by using ANOVA; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 136.62, 90% CI 2-sided [103.20 to 180.87]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of Talazoparib: Alone and in Combination With Rifampin
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 15
hr*pg/mL | 196631.34 (32) | 196100.69 (33)
Statistical Analysis 1: Comparison: Talazoparib 1.0 mg Alone vs Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 105.37, 90% CI 2-sided [98.04 to 113.24]

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of Talazoparib: Alone and in Combination With Rifampin
Description: as for outcome 4
Time Frame: as for outcome 4
Population: PK analysis population included all participants who enrolled, treated and had at least 1 of the talazoparib PK parameters. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 12
hr*pg/mL | 209521.62 (34) | 194307.67 (36)
Statistical Analysis 1: Comparison: Talazoparib 1.0 mg Alone vs Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric LS Mean Ratio = 102.04, 90% CI 2-sided [94.02 to 110.74]

7. Secondary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Talazoparib: Alone and in Combination With Itraconazole
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 19 | 15
Hours | 1.00 [0.5 to 24.1] | 1.02 [0.5 to 4.0]

8. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Talazoparib: Alone and in Combination With Itraconazole
Description: Terminal elimination half-life was defined as time measured for the plasma concentration of talazoparib to decrease by one half. T1= Time frame for "Talazoparib 0.5 mg Alone" and T2= time frame for "Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID".
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 18 | 12
Hours | 101.26 (26.315) | 118.47 (23.600)

9. Secondary Outcome: Apparent Clearance (CL/F) of Talazoparib: Alone and in Combination With Itraconazole
Description: Clearance of talazoparib was measure of the rate at which it was metabolized or eliminated by normal biological processes. T1= Time frame for "Talazoparib 0.5 mg Alone" and T2= time frame for "Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID".
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 18 | 12
Liter per hour | 4.55 (42) | 3.29 (36)

10. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Talazoparib: Alone and in Combination With Itraconazole
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of talazoparib would need to be uniformly distributed to produce its desired plasma concentration. T1= Time frame for "Talazoparib 0.5 mg Alone" and T2= time frame for "Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID".
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Talazoparib 0.5 mg Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID
Number analyzed (Participants) | 18 | 12
Liter | 644.81 (42) | 552.01 (27)

11. Secondary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Talazoparib: Alone and in Combination With Rifampin
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 15
Hours | 1.00 [0.5 to 24.0] | 1.00 [0.5 to 8.0]

12. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Talazoparib: Alone and in Combination With Rifampin
Description: Terminal elimination half-life was defined as time measured for the plasma concentration of talazoparib to decrease by one half. T3= Time frame for "Talazoparib 1.0 mg Alone" and T4= time frame for "Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD".
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 12
Hours | 92.05 (17.679) | 80.61 (16.540)

13. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Talazoparib: Alone and in Combination With Rifampin
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of talazoparib would need to be uniformly distributed to produce its desired plasma concentration. T3= Time frame for "Talazoparib 1.0 mg Alone" and T4= time frame for "Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD".
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 12
Liter | 623.89 (30) | 588.14 (33)

14. Secondary Outcome: Apparent Clearance (CL/F) of Talazoparib: Alone and in Combination With Rifampin
Description: Clearance of talazoparib was measure of the rate at which it was metabolized or eliminated by normal biological processes. T3= Time frame for "Talazoparib 1.0 mg Alone" and T4= time frame for "Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD".
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Talazoparib 1.0 mg Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 17 | 12
Liter per hour | 4.77 (34) | 5.15 (36)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. A TEAE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to end of study (up to 61 days)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib. Here, 1 participant received 2 doses of rifampin and the SAE anastomotic stenosis took place in the "rifampin" period. Originally, this SAE was attributed to the "talazoparib only" period under the assumption that the participant did not receive any dose of rifampin. This SAE was shifted from the "talazoparib only" period to the "rifampin" period.
Measure: Count of Participants; unit: Participants
Groups:
- Itraconazole 100 mg BID Alone: Participants those who had received single oral dose of talazoparib 0.5 mg on Day 1 in Period 1, received oral dose of itraconazole 200 mg (100 mg BID) from Day 16 to Day 22 in Period 2.
- Rifampin 600 mg QD Alone: Participants those who had received a single oral dose of talazoparib 1.0 mg on Day 1 in Period 1, received oral dose of rifampin 600 mg QD from Day 16 to Day 24 in Period 2.
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg Alone | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 19 | 16 | 15 | 17 | 17 | 15
Participants
  AEs | 12 | 3 | 5 | 6 | 9 | 5
  SAEs | 3 | 0 | 1 | 0 | 2 | 0

16. Secondary Outcome: Number of Participants With Clinical Significance Abnormalities in Laboratory Parameters
Description: Chemistry:(sodium135-146,potassium3.5-5.5,chloride95-109,glucose3.3-5.5,urea2.8-7.2,calcium2.2-2.65,phosphate0.8-1.45,triglyceride0.4-1.7,cholesterol2.6-5.2)millimoles/L, (bilirubin[direct0-3,total2-21],creatinine53- 110)micromole/L, (albumin35-52,protein65-83)g/L,(alkaline phosphatase30-120, aspartate amino[A]transferase[T]4-46, alanine AT4-49, lactic acid dehydrogenase200-460, gammaglutamylT7-50,creatinine kinase24-170)U/L. Hematology: hemoglobin(Hb)120-177, hematocrit0.35-0.49L/L, RBC4-5.9T/L, (platelet150- 400,WBC4-10,basophil<0.10,eosinophil<0.40, neutrophil1.50-7.00,monocyte<1.20,lymphocyte1.0 -3.70)G/L. Urine:(glucose,protein,ketone,Hb:negative/positive), specific gravity1.010-1.030g/cm^3, pH4.8-7.8, pale yellow-deep amber, microscopy[WBC0-5,leukocyte0-5,Hb0-3,cast0-1,bacteria0-500,epithelial0-6])Pcs/area. Coagulation:(activated partial thromboplastine time25-43,prothrombin time13.7-15.6) seconds,international normalized ratio0.89-1.1. Investigator judged clinical significance.
Time Frame: Baseline up to end of study (up to 61 days)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg Alone | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 19 | 16 | 15 | 17 | 17 | 15
Participants | 3 | 0 | 1 | 2 | 1 | 1

17. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign abnormalities: a) systolic blood pressure (SBP): 1) minimum less than (<) 90 millimeter of mercury (mmHg), 2) change from baseline maximum decrease greater than equal to (>=) 30 mmHg, 3) change from baseline maximum increase >=30 mmHg; b) diastolic blood pressure (DBP): 1) minimum <50 mmHg, 2) change from baseline maximum decrease >=20 mmHg, 3) change from baseline maximum increase >=20 mmHg; c) supine pulse rate: 1) minimum <40 beats per minute (bpm), 2) maximum >120 bpm; d) standing pulse rate: 1) minimum <40 bpm and 2) maximum >140 bpm. Clinical significance of vital signs abnormalities was judged by investigator.
Time Frame: Baseline up to end of study (up to 61 days)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg Alone | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 19 | 16 | 15 | 17 | 17 | 15
Participants | 0 | 0 | 1 | 0 | 0 | 1

18. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: ECG abnormalities: a) QT Interval: new absolute values greater than (>) 450, >480, >500 milliseconds (msec), increase from baseline >30 and >60 msec, b) QT interval using Fridericia's correction (QTcF) Interval: new absolute values >450, >480, >500 msec, increase from baseline >30 and > 60 msec, c) Heart rate: increase from baseline >25 percentage (%) and to a value >100 bpm, decrease from baseline >25% and to a value <50 bpm, d) PR Interval: increase from baseline > 25% and to a value >200 msec, e) QRS duration: increase from baseline > 25% and to a value >100 msec. Clinical significance of ECG abnormalities was judged by investigator.
Time Frame: Baseline up to end of study (up to 61 days)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg Alone | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 19 | 16 | 15 | 17 | 17 | 15
Participants | 0 | 1 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included examination of abdomen, cardiovascular, eyes, ears, nose, throat, general appearance, head, neck, thyroid, lymph nodes, musculoskeletal, neurological, skin / subcutaneous tissue, thorax / lungs, abdomen including spleen size, breasts (female only) and respiratory. Clinical significance of physical examination was judged by investigator.
Time Frame: Baseline up to end of study (up to 61 days)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg Alone | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
Number analyzed (Participants) | 19 | 16 | 15 | 17 | 17 | 15
Participants | 0 | 0 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to 61 days)
Description: One participant received 2 doses of rifampin and the SAE anastomotic stenosis took place in the "rifampin" period. Originally, this SAE was attributed to the "talazoparib only" period under the assumption that the participant did not receive any dose of rifampin. This SAE was shifted from the "talazoparib only" period to the "rifampin" period.
Groups:
- Talazoparib 1.0 mg: Participant received a single oral dose of talazoparib 1.0 mg on Day 1 followed by washout of 14 days in Period 1.
Arm/Group | Talazoparib 0.5 mg Alone | Itraconazole 100 mg BID Alone | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID | Talazoparib 1.0 mg | Rifampin 600 mg QD Alone | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/16 | 1/15 | 0/17 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/19 | 0/16 | 1/15 | 0/17 | 2/17 | 0/15
Other Adverse Events (participants affected / at risk) | 12/19 | 3/16 | 5/15 | 6/17 | 9/17 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 0.5 mg Alone (N=19) | Itraconazole 100 mg BID Alone (N=16) | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID (N=15) | Talazoparib 1.0 mg (N=17) | Rifampin 600 mg QD Alone (N=17) | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD (N=15)
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 0.5 mg Alone (N=19) | Itraconazole 100 mg BID Alone (N=16) | Talazoparib 0.5 mg in Combination With Itraconazole 100 mg BID (N=15) | Talazoparib 1.0 mg (N=17) | Rifampin 600 mg QD Alone (N=17) | Talazoparib 1.0 mg in Combination With Rifampin 600 mg QD (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In this study 1 participant received 2 doses of rifampin and the SAE anastomotic stenosis took place in the "rifampin" period. Originally, this SAE was attributed to the "talazoparib only" period under the assumption that the participant did not receive any dose of rifampin. This SAE was shifted from the "talazoparib only" period to the "rifampin" period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results

DOCUMENTS (2):
  • Study Protocol (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03077607/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03077607/SAP_000.pdf